CLINICAL TRIAL: NCT06056960
Title: Preventing the Progression of Physical Disability and Promoting Brain Functional Adaptation in People With Multiple Sclerosis: Integration of Early Rehabilitative Treatment and Multimodal Clinical and Instrumental Assessment - Part B
Brief Title: Preventing the Progression of Multiple Sclerosis: Early Rehabilitative Treatment and Multimodal Assessment - Part B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: IRCCS San Raffaele (Other); Azienda Sanitaria Locale di Cagliari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 03_17/02/2021 Part B
Record Dates: First submitted 2023-09-11; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
Keywords: early phase; non-disabled
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): The experimental group will perform a combination of endurance and balance training tailored to the subject.
  Interventions: Other: Tailored Physical Activity
- Usual Activity (No Intervention): The control group will perform their usual daily activities.

INTERVENTIONS:
Other: Tailored Physical Activity — The intervention will comprise 16 sessions (2 sessions/week). 30 minutes of walking training wearing a heart rate (HR) monitor to keep exercise intensity below 70% of maximal HR.
  Right after, 30 minutes of balance exercises will be performed. An experienced physical therapist will tailor exercises. Subjects will be taught how to perform the exercises by themselves. A booklet will be provided to provide guidelines. A physical therapist will call subjects, every training day to check for any problem.
  Arms: Physical Activity

SUMMARY:
It is widely recognized that physical exercise is safe and people with moderate Multiple Sclerosis (MS) are encouraged to train regularly to improve their skills in motor task execution. Several studies demonstrated that these activities represent an effective low-cost therapy which leads to significant and clinically meaningful improvements in gait and balance in people with MS (PwMS) with mild to moderate walking dysfunction, possibly also by promoting brain plasticity.

There is general agreement within the scientific community on the importance of timing intervention also during the early stages of MS to preserve or improve walking and balance abilities and fostering brain functional adaptation, thus slowing down the disease progression. Previous studies highlighted the need to early identify and manage gait disorders using a multimodal approach tailored on individual's need. Moreover, Functional Near-Infrared Spectroscopy (fNIRS) measures blood flow which accompanies neuronal activity and thus, it can provide spatial information about changes in cortical activation patterns due to the possible effects of exercise on cortical plasticity.

To the best of the investigators knowledge, no published studies have assessed the effect of exercise on mobility and brain activity in PwMS with minimal or clinically undetectable disability. This emphasizes the need of trials investigating the effect of walking exercise as preventive strategy on MS clinical worsening.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years
* Stable disease course (without worsening over 1 point at the Expanded Disability Status Scale in the last 3 months)

Exclusion Criteria:

* Major depression
* Mini-Mental State Examination < 27
* Other cardiovascular or orthopedic diseases that interfere with physical exercise
* Progressive course of the disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale (FSS) | Baseline, Post, FollowUp_6month
  Is a 9-item self-administered questionnaire to measure the perceived impact of fatigue. The minimum score is 9 and maximum score possible is 63. Higher scores represent greater fatigue severity. If the score is calculated as the mean score of the 9 items, the cut-off score for the presence of the symptom fatigue is set as scores higher than 4.

SECONDARY OUTCOMES:
Differences in oxygenated hemoglobin (Delta oxyHb) | Baseline, Post, FollowUp_6month
  The differences in oxyHb during task period and resting state. Data will be extracted from functional Near InfraRed Spectroscopy (fNIRS) assessment.
Six Minute walking test (6MWT) | Baseline, Post, FollowUp_6month
  Gait asymmetry and regularity extracted from Inertial Measurement Unit's during the six minute walking test.
Number of steps/day | Baseline, Post, FollowUp_6month
  Assessed by activity trackers, a non-invasive method of monitoring human rest/activity cycles. Subjects will be monitored for 1 week wearing an actigraph.
Endurance walking capacity | Baseline, Post, FollowUp_6month
  Assessed as the distance walked over 6 minutes as a sub-maximal test of endurance (6MWT).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Rovaris, MD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi; Raffaella Chieffo, MD, Principal Investigator — IRCCS Ospedale San Raffaele; Eleonora Cocco, MD, Principal Investigator — Ospedale Binaghi ASL Cagliari, Sardegna
Locations (3):
- Italy (3):
  - Ospedale Binaghi ASL Cagliari, Cagliari
  - IRCCS Ospedale San Raffele, Milan
  - IRCCS Fondazione Don Carlo Gnocchi, Milan